CLINICAL TRIAL: NCT03940313
Title: Biotensegrity: Thoracolumbar Fascial Integrity in Chronic Low Back Pain
Status: Completed | Type: Observational
Sponsor: ProloAustin (Other)
Responsible Party: Principal Investigator, Bradley D. Fullerton, MD, Adjunct Assistant Professor, Texas A&M College of Medicine, ProloAustin
Other Study IDs: ICMS-2019-004
Record Dates: First submitted 2019-05-04; First posted 2019-05-07 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Musculoskeletal Pain; Low Back Pain; Myofascial Pain
Keywords: Chronic Low Back Pain; Myofascial pain; Tensegrity; Prolotherapy; Platelet-Rich Plasma
MeSH Terms: conditions — Musculoskeletal Pain; Low Back Pain | interventions — Prolotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects: Participants >18 years old who meet inclusion and exclusion criteria, and have findings on physical exam and ultrasound that suggest potential benefit from prolotherapy.
  Interventions: Procedure: Prolotherapy
- Controls: Participants >or =18 years old who do not complain of lower back pain, but consent to have physical examination testing and musculoskeletal ultrasound of the lower back to evaluate these areas.

INTERVENTIONS:
Procedure: Prolotherapy — Musculoskeletal injection of lidocaine + 15% dextrose into damaged tissue
  Other Names: injection therapy
  Groups: Subjects

SUMMARY:
This is a prospective study on chronic low back pain patients aimed at investigating how findings on a physical examination and musculoskeletal ultrasound may correlate with myofascial damage in the lower back. By comparing these findings with a control group and collecting follow up data on patients treated in the course of normal clinical practice, the investigators will be able to discern if fascial pathology contributes to chronic low back pain and if this treatment approach may provide clinical benefit to patients in the form of pain reduction and/or reduction in pain medication use.

DETAILED DESCRIPTION:
This is a prospective, observational clinical study that will be run through a private practice clinic.

New patients to the clinic that complain of chronic lower back pain will be evaluated for inclusion and exclusion criteria and appropriately recruited and enrolled into the study. The baseline evaluation will take approximately 1.5hours to complete, and will include the following: a standardized pain scale questionnaire; a baseline questionnaire that assesses duration of current pain and previous interventions; physical examination with novel techniques to assess strength; and musculoskeletal ultrasound in the lower back.

Specific physical examination techniques will assess strength of the subject on both prone straight leg raise as well as hip external rotation. Then, the investigators will test how adding myofascial tension along the lower back may affect these results. Musculoskeletal ultrasound will examine specifically the aponeurosis of the erector spinae and the posterior layer of the thoracolumbar fascia at T11, T12, and L1. These areas will be graded on a 4-point scale (0 to 3), evaluating compressibility and heterogeneity of the tissue.

Participants who have myofascial damage identified on ultrasound and are scheduled for injection treatment as part of normal clinical care will have a diagnostic injection of prolotherapy (0.3% lidocaine + 15% dextrose) in those areas as the first step of the procedure. Pre and post injection muscle testing will be performed. The treatment session then will be completed per normal clinical care; this may include injection at other locations and injection of autologous platelet-rich plasma. Routine follow-up will be scheduled at 3 months.

At 3 months, the follow-up visit will include the following: the same pain scale questionnaire; a follow-up questionnaire to assess changes in function and pain medication; physical examination as before; musculoskeletal ultrasound in the specified areas.

New patients to the clinic who do not have chronic low back pain >12 weeks will be asked to participate as controls, and will undergo a similar questionnaire, and the same physical examination and musculoskeletal ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 18 years old
* Chronic lower back pain > or = 12 weeks duration

Exclusion Criteria:

* History of stroke preventing bilateral muscle strength testing
* History of scoliosis that may affect myofascial dynamics
* Acute radiculopathy/sciatica or pain that limits movement for physical examination
* Unable to lie prone for physical examination

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with chronic lower back pain that meet inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
Pain Scale | At baseline and at 3 month follow-up.
  Improved lower back pain / functionality.
  Pain will be discerned on a scale from 0 to 10, with 0 being no pain and 10 being the worst pain the participant has experienced. There will be no subscales provided, and only whole numbers will be allowed to be reported.
MSK Ultrasound | At baseline and at 3 month follow-up
  Musculoskeletal ultrasound will evaluate specific areas in the lower back on a 4-point scale (0 to 3), evaluating compressibility and heterogeneity of the tissue. The scale is described as follows:
  0= No significant compressibility (well defined)
  1. Mild compressibility but no translation (heterogeneous)
  2. Moderate compressibility, mild translation (heterogeneous, poorly organized)
  3. Significant compressibility and translation (heterogeneous, poorly organized)
  The results from each of the areas evaluated will then be summed for a total composite score. All values, including the individual area score and total composite score, will be recorded. Higher scores are considered worse outcomes. The results of the ultrasound evaluation will be determined solely by the principal investigator.

SECONDARY OUTCOMES:
Medications | At baseline and at 3 month follow-up
  Reduced use (dose or frequency) of pain medications

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Fullerton, MD, Principal Investigator — ProloAustin
Locations (1):
- ProloAustin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dischiavi SL, Wright AA, Hegedus EJ, Bleakley CM. Biotensegrity and myofascial chains: A global approach to an integrated kinetic chain. Med Hypotheses. 2018 Jan;110:90-96. doi: 10.1016/j.mehy.2017.11.008. Epub 2017 Nov 20. PMID 29317079
- [Background] Swanson RL 2nd. Biotensegrity: a unifying theory of biological architecture with applications to osteopathic practice, education, and research--a review and analysis. J Am Osteopath Assoc. 2013 Jan;113(1):34-52. doi: 10.7556/jaoa.2013.113.1.34. PMID 23329804
- [Background] Fullerton BD, Reeves KD. Ultrasonography in regenerative injection (prolotherapy) using dextrose, platelet-rich plasma, and other injectants. Phys Med Rehabil Clin N Am. 2010 Aug;21(3):585-605. doi: 10.1016/j.pmr.2010.06.003. PMID 20797551
- [Background] Todorov PT, Nestorova R, Batalov A. Diagnostic value of musculoskeletal ultrasound in patients with low back pain - a review of the literature. Med Ultrason. 2018 Feb 4;1(1):80-87. doi: 10.11152/mu-1245. PMID 29400373
- See also: Clinical facility for study — https://proloaustin.com/